CLINICAL TRIAL: NCT06145971
Title: Assessing the Impact of Brief Cognitive Behavioural Therapy for Insomnia on Sleep Difficulties in a Dissociative Seizure Population, Using a Single-Case Experimental Design.
Brief Title: Assessing the Impact of Brief CBTi on Dissociative Seizures: SCED
Acronym: CBTi 4 DS:SCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: William Quarriers Scottish Epilepsy Centre (Unknown)
Responsible Party: Principal Investigator, Sarah Adam, Trainee Clinical Psychologist, Post-Graduate Researcher, University of Glasgow
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331958; 331958 (Other: Integrated Research Application System)
Record Dates: First submitted 2023-11-10; First posted 2023-11-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Dissociative Seizures; Functional Seizures; Psychogenic Nonepileptic Seizures; Insomnia; Dissociation; Sleep Disorder
Keywords: dissociative seizures; SCED; insomnia; functional seizures; psychogenic nonepileptic seizures; sleep disorder; dissociation
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Sleep Initiation and Maintenance Disorders; Dissociative Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (SCED) methodology using multiple baseline across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline phase (No Intervention): Randomly allocated baseline phase (no intervention) of 5, 7, or 9 days.
- Intervention - bCBTi (Experimental): Two sessions of brief Cognitive Behavioural Therapy for insomnia (bCBTi). This will involve a clinical psychologist meeting with the participant for two sessions, three days apart, to provide bCBTi, which will involve a cognitive and a behavioural therapy technique.
  Interventions: Behavioral: brief Cognitive Behavioural Therapy for Insomnia (bCBTi)

INTERVENTIONS:
Behavioral: brief Cognitive Behavioural Therapy for Insomnia (bCBTi) — Two sessions of Cognitive Behavioural Therapy for Insomnia, encompassing a cognitive therapy technique and a behavioural technique as a minimum.
  Arms: Intervention - bCBTi

SUMMARY:
Some people experience a temporary change in behaviour and consciousness, that often involves a collapse and/or shaking limb movements. These are referred to as 'Dissociative seizures'. Those who experience such seizures have been found to also display high levels of dissociation, which can be described as a change in your conscious experience and may include gaps in your memory for events. It is thought that people who experience dissociative seizures also often have difficulties with their sleep. Having difficulties with sleep may make these seizures and the amount of dissociation an individual experiences worse. Greater dissociation may be additionally linked to worsening dissociative seizures. A psychological treatment for sleep difficulties called Cognitive Behavioural Therapy for Insomnia (CBTi), has been found to be effective in reducing sleep difficulties.

The main questions this study aims to answer are:

1. Does brief CBTi (bCBTi) improve sleep difficulties in those with dissociative seizures?
2. Does bCBTi reduce the frequency of dissociative seizures?
3. Does bCBTi reduce self-reported levels of dissociation in participants?
4. Does improving sleep difficulties lead to improvements in quality of life, mood and anxiety levels?
5. Is bCBTi a feasible intervention to administer in an inpatient setting?

This study will investigate whether improving sleep by administering a brief version of CBTi leads to an improvement in levels of dissociation and dissociative seizure frequency. It will also investigate whether brief CBTi is a feasible treatment method for sleep difficulties in an inpatient setting.

Participants who have dissociative seizures and sleep difficulties that could be diagnosed as insomnia will be randomly assigned to a baseline phase of 5, 7 or 9 days, where they will fill out daily questionnaires on their sleep, dissociation and number of seizures. They will then begin a 10-day intervention phase where they will attend two sessions of brief CBTi, whilst also completing daily measures. This will allow us to see whether their scores on the sleep and dissociation measures improve when the intervention begins. Participants will be asked to wear an Actiwatch during the night, to gather information on their movement levels during the night. Information on changes in quality of life, mood and anxiety levels following the sleep intervention will also be collected.

DETAILED DESCRIPTION:
Design: This study will use a Multiple Baseline Single Case Experimental Design (SCED). This design has been chosen as it can test the effectiveness of an intervention on a small number of participants. This is of benefit as it allows the piloting of a novel intervention, which brief Cognitive Behavioural Therapy for Insomnia (bCBTi) for those with dissociative seizures will be. It will involve each participant being randomly assigned to a baseline phase of three possible lengths: 5 days, 7 days and 9 days. This will be done using https://www.randomizer.org/ which will generate a random order of the three categories. During the baseline phase, sleep difficulties and levels of dissociation will be measured on a daily basis. The participant will then begin the intervention phase, where they will receive two sessions of bCBTi. Sleep difficulties and levels of dissociation will continue to be measured on a daily basis during the intervention phase. Participants can therefore serve as their own controls. The multiple baseline element controls for time as a confounding variable which increases the study's internal validity, and allows the relationship between variables to be viewed as causal rather than correlational. Guidelines for constructing good quality SCEDs have been used to inform the study protocol.

Recruitment: The study will take place at the William Quarrier Scottish Epilepsy Centre (WQSEC), recruiting current inpatients who meet the criteria for inclusion in the study. Potential participants will be identified and approached initially by the clinical nurse specialist (CNS) on the ward who has access to patient information and is alerted of any new inpatients. The CNS will provide the potential participant with an information sheet, and ask if they would consent to the principal investigator speaking to them to go through it, answer any questions and obtain informed consent. If the participant agrees to participating, the baseline measures will also be completed at this stage. Overall, the recruitment stage should take around 1 hour of participant's time over a couple of days.

Baseline phase: The participant will then enter a randomly assigned baseline phase of 5, 7 or 9 days in length, which will involve them completing two short measures on a daily basis and wearing an actiwatch during the night. It will take around 10-15 minutes to complete the measures each day. Nursing and/or Health Care Assistants on the ward may assist with prompting participants to complete the measures throughout the duration of the study if they have capacity in addition to their primary clinical duties.

Intervention phase: Once they have completed their baseline phase, they will begin the intervention phase, which will involve attending two sessions of bCBTi with a clinical psychologist on the ward. Each session will last between an hour to an hour and a half. The sessions will be three days apart, one on a Monday and one on a Friday. The participants will continue to complete daily measures during this time, and will continue to wear the actiwatches.

Post-intervention phase and study completion: Following the two sessions of bCBTi, the participants will continue to complete the daily measures and wear the actiwatch for 7 days. Following this, the principal investigator will meet with the participants to complete the post intervention measures, which are the same as the pre-intervention measures. At this meeting, the principal investigator will also debrief the participants on the study. This meeting will take around an hour.

ELIGIBILITY:
Inclusion Criteria:

* aged 18+ (no upper age limit);
* can speak and read English fluently;
* must score ≤16 on the Sleep Conditions Indicator (SCI);
* must demonstrate compelling evidence that at least some of their seizures are likely to be dissociative, based on at least one of the following:

  1) Opinion of the referring consultant, WQSEC consultant, or WQSEC clinical nurse specialist, based on:
* Direct witnessing of seizure(s)
* Review of video footage
* Semiology as suggested by reliable patient or family history. 2)EEG assessment showing seizures without EEG change correlated. The participant must have received feedback that they are experiencing dissociative seizures and is accepting of this as an explanation.

Exclusion Criteria:

* active and significant mental health problems and/or moderate to severe learning disabilities (IQ score of ≤50);
* unable to give informed consent;
* non-fluent English speakers;
* current participation in another research study;
* dissociative seizures that have been assessed by the WQSEC clinical psychologist and/or consultant as potentially deliberate behaviour driven by secondary gain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | Measured daily, from baseline to final day of post-intervention phase (day 1 up to day 21).
  Total time spent asleep in bed in minutes. Measured using actigraphy and a sleep diary completed by the participant. Higher scores indicated longer time spent asleep.
Wake after sleep onset (WASO) | Measured daily, from baseline to final day of post-intervention phase (day 1 up to day 21).
  Total time spent awake after sleep onset in minutes. Measured using actigraphy and a sleep diary completed by the participant. Higher scores indicate longer time spent awake.
Number of night time awakenings | Measured daily, from baseline to final day of post-intervention phase (day 1 up to day 21).
  Total number of awakenings during the night. Measured using actigraphy and a sleep diary completed by the participant. Min = 0 - no Max. Lower scores indicate fewer night time awakenings.
Sleep onset latency (SOL) | Measured daily, from baseline to final day of post-intervention phase (day 1 up to day 21).
  Time taken to fall asleep in minutes measured using actigraphy and a sleep diary completed by the participant. Higher scores indicate greater SOL.

SECONDARY OUTCOMES:
Time in bed (TIB) | Measured daily, from baseline to final day of post-intervention phase (day 1 up to day 21).
  Total time spent in bed in minutes with higher scores indicating longer time spent in bed. Measured using a sleep diary completed by the participant.
Insomnia Classification | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  Sleep Condition Indicator (SCI) score. Min score= 0 - Max= 32 with lower scores indicating poorer sleep.
Anxiety symptoms | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  Generalized Anxiety Disorder Questionnaire (GAD-7) score. Min= 0 - Max= 21 with higher scores indicating more severe symptoms.
Depressive symptoms | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E). 6-item self-report questionnaire, min = 6, max = 24. Greater scores indicate more severe symptoms.
Attendance | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  Attendance of bCBTi sessions. Min = 1, max = 2.
Quality of Life | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  Patient Weighted Quality of Life in Epilepsy (QoLIE-10-P). Min = 10, max = 51 with greater scores indicating lower quality of life.
Dissociation | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  Dissociative Experiences Scale-II (DES-II), a 28-item questionnaire where items are measured on the percentage of time each item is experienced (0-100%). Scores ≥30 indicate the presence of a dissociative disorder.
Daily dissociation | Measured at day 1 and again at the end of the post-intervention phase, day 17-21.
  The Clinician-Administered Dissociative States Scale-6 (CADSS-6). Min = 6, max = 24, with greater scores indicating greater levels of dissociation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jessica Fish, BSc, PhD, DClinPsy, Study Director — University of Glasgow
Locations (1):
- William Quarrier Scottish Epilepsy Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD.

REFERENCES:
- [Background] Mousa S, Latchford G, Weighall A, Nash H, Murray-Leslie R, Reuber M, Relton SD, Graham CD. Evidence of objective sleep impairment in nonepileptic attack disorder: A naturalistic prospective controlled study using actigraphy and daily sleep diaries over six nights. Epilepsy Behav. 2021 Apr;117:107867. doi: 10.1016/j.yebeh.2021.107867. Epub 2021 Mar 5. PMID 33684785
- [Background] Brown RJ, Reuber M. Psychological and psychiatric aspects of psychogenic non-epileptic seizures (PNES): A systematic review. Clin Psychol Rev. 2016 Apr;45:157-82. doi: 10.1016/j.cpr.2016.01.003. Epub 2016 Mar 16. PMID 27084446
- [Background] Campbell MC, Smakowski A, Rojas-Aguiluz M, Goldstein LH, Cardena E, Nicholson TR, Reinders AATS, Pick S. Dissociation and its biological and clinical associations in functional neurological disorder: systematic review and meta-analysis. BJPsych Open. 2022 Dec 1;9(1):e2. doi: 10.1192/bjo.2022.597. PMID 36451595